CLINICAL TRIAL: NCT01347983
Title: Extension Study of Tocilizumab Long Term Treatment of Moderate to Severe Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharma Taiwan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA230TW EX
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tocilizumab+Methotrexate(MTX) — Tocilizumab: 8 mg/kg every 4 weeks, IV infusion Methotrexate: 10-20 mg/week

SUMMARY:
24 week open-labeled extension study to continue monitoring the same group of patients in the previous MRA230TW phase IIIb trial in order to evaluate the long term efficacy and safety of tocilizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had completed at least 5 out of the 7 visits scheduled for weeks 2, 4, 8, 12, 16, 20 and 24 in the tocilizumab Phase IIIb study(MRA230TW).
* Patients assigned in the Phase IIIb study(MRA230TW), who had received scheduled dose for at least 16 weeks but still failed to achieve adequate treatment response characterized by ACR20

Exclusion Criteria:

* Patients who have received a major surgery including joint surgery 8 weeks prior to the screening or are scheduled to be operated within 6 months after the enrolment.
* Patients with rheumatoid autoimmune disease other than RA, including but not limited to SLE(system lupus erythematosus), or significant systemic involvement secondary to RA.
* Patients who belong to the Class IV of the ACR classification criteria for functional status of RA. (ACR Amended Criteria for the Classification of Functional Capacity in Rheumatoid Arthritis; Class IV: Largely or wholly incapacitated with patient bedridden or confined to wheel chair, permitting little or no self-care).
* Patients with a history of hypersensitivity to human, humanized or murine monoclonal antibodies or patients with contraindication for them.
* Patients who currently have or have a history of recurrence of bacterial, viral,fungal, or mycobacterial infections or other infectious diseases; tuberculosis(TB),atypical mycobacterial disease, clinically significant granulomatous disease on chest radiograph, hepatitis B, hepatitis C, or herpes zoster and etc. However, a patient with hand & foot fungal infections can participate.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an American College of Rheumatology 70 (ACR70) response | at week 24

SECONDARY OUTCOMES:
Proportion of patients with ACR50 response | at week 24
Proportion of patients with ACR20 response | at week 24
Mean change from baseline of Swollen joint count(SJC) and Tender joint count(TJC) respectively | at baseline and week 24
Mean change from baseline in disease activity using 28-joint modified disease activity score (DAS28) | at baseline and week 24
Proportion of patients achieving DAS28 remission (DAS28 < 2.6) | at week 24
Adverse event incidence | from baseline to week 24
Mean change from baseline to evaluation visits in vital signs | from baseline to week 24
Change in Electrocardiogram. From baseline to evaluation visits | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative hematological exam results. | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative Biochemical exam of blood results. | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative serum lipid exam results. | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative urinalysis results. | from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiaki Someya, Study Chair — Chugai Pharma Taiwan
Locations (12):
- Taiwan (12):
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Memorial Hospital -Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District